CLINICAL TRIAL: NCT06871332
Title: The Effect of Progressive Relaxation Exercise on Pain, Anxiety and Patient Satisfaction Related to Femoral Sheath Removal: a Randomized Controlled Study
Brief Title: Progressive Relaxation Exercise on Pain, Anxiety and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof.Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/543
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Effect of Progressive Relaxation Exercise
Keywords: Anxiety; Femoral Sheath; Pain; Progressive Relaxation Exercise; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive relaxation exercises group (Experimental): Patients in the intervention group performed progressive relaxation exercise for 20 minutes before femoral sheath removal.
  Interventions: Other: Progressive relaxation exercise group
- Control group (No Intervention): The patients in the control group received the standard practice of the clinic.

INTERVENTIONS:
Other: Progressive relaxation exercise group — Patients in the intervention group performed progressive relaxation exercise for 20 minutes before femoral sheath removal.
  Arms: Progressive relaxation exercises group

SUMMARY:
This single-center, prospective, randomized controlled trial was completed with a total of 70 patients, 35 in each of the intervention and control groups. Data were collected using the Patient Information Form, Visual Analogy Scale and State-Trait Anxiety Inventory. Patients in the intervention group performed progressive relaxation exercise for 20 minutes before femoral sheath removal. The patients in the control group received the standard practice of the clinic.

DETAILED DESCRIPTION:
This study aimed to determine the effect of progressive relaxation exercise (PRE) applied to patients undergoing percutaneous coronary intervention (PCI) on pain, anxiety and patient satisfaction related to femoral sheath removal. This single-center, prospective, randomized controlled trial was completed with a total of 70 patients, 35 in each of the intervention and control groups. Data were collected using the Patient Information Form, Visual Analogy Scale and State-Trait Anxiety Inventory. Patients in the intervention group performed PRE for 20 minutes before femoral sheath removal. The patients in the control group received the standard practice of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* able to speak and understand Turkish,
* over 18 years of age,
* intervened in the femoral region,
* with only one catheter in the femoral region,
* without vision and hearing problems,
* undergoing angiography procedure for the first time,
* with normal vital signs,
* who have not been administered analgesics for any reason prior to sheath removal after the procedure,
* patients who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* patients with chronic pain using transdermal patches,
* patients with impaired time and place orientation,
* patients with psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Pain level | One minute after femoral sheath removal
  Patients' pain is evaluated with the Visual Analog Scale (VAS) .The VAS is a 10 cm long ruler drawn horizontally or vertically. Patients were told that 0 on the scale means no pain and 10 means unbearable pain at the highest level. The patient was asked to mark the point on this scale indicating the level of pain they felt.
Anxiety level | One minute after femoral sheath removal
  Patients' anxiety is evaluated with the Visual Analog Scale (VAS). The VAS is a 10 cm long ruler drawn horizontally or vertically. patients were told that 0 on the scale means no anxiety and 10 means unbearable anxiety at the highest level. The patient was asked to mark the point on this scale indicating the level of anxiety they felt.
Patient satisfaction | One minute after sheath removal
  Patients' anxiety is evaluated with the Visual Analog Scale (VAS). The VAS is a 10 cm long ruler drawn horizontally or vertically. It was explained to the patient that the number 0 indicated no satisfaction with the application and the number 10 indicated the highest level of satisfaction and the patient was asked to mark on the ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No